CLINICAL TRIAL: NCT07246070
Title: The Efficacy and Safety of Nano-crystalline Megestrol Acetate for the Prevention of Nausea and Vomiting Caused by Emetogenic Chemotherapy: a Randomized, Controlled, Multicenter Clinical Study
Brief Title: Nano-crystalline Megestrol Acetate for Chemotherapy-induced Nausea and Vomiting
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AIPING ZHOU (Other)
Collaborators: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor-Investigator, AIPING ZHOU, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCC5420
Record Dates: First submitted 2025-09-16; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting (CINV)
MeSH Terms: conditions — Vomiting | interventions — Ondansetron

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single-arm study group (Experimental)
  Interventions: Drug: nanocrystalline megestrol acetate combined with ondansetron
- nanocrystalline megestrol acetate group (Experimental)
  Interventions: Drug: nanocrystalline megestrol acetate combined with ondansetron
- dexamethasone group (Active Comparator)
  Interventions: Drug: dexamethasone combined with ondansetron

INTERVENTIONS:
Drug: nanocrystalline megestrol acetate combined with ondansetron — nanocrystalline megestrol acetate (5 ml PO, qd, Day 1-Day 14), ondansetron (8 mg IV, qd, Day 1).
  Arms: Single-arm study group; nanocrystalline megestrol acetate group
Drug: dexamethasone combined with ondansetron — dexamethasone (8 mg IV, qd, Day 1), ondansetron (8 mg IV, qd, Day 1)
  Arms: dexamethasone group

SUMMARY:
The primary objective of this clinical study is to evaluate the efficacy and safety of nanocrystalline megestrol acetate combined with a 5-HT3 receptor antagonist for the prophylaxis of nausea and vomiting caused by moderately emetogenic chemotherapy drugs.

The study population consists of gastric adenocarcinoma patients who are scheduled to receive their first course of moderately emetogenic chemotherapy (PD-1/PD-L1 immune checkpoint inhibitors combined with the CAPOX regimen). This study is divided into two phases. The first phase is a single-arm study design, with the primary objective of preliminarily assessing the efficacy and safety of nanocrystalline megestrol acetate combined with a 5-HT3 receptor antagonist for the full-course management of nausea and vomiting caused by moderately emetogenic chemotherapy drugs. The second phase will adopt a randomized, controlled, multicenter trial design. Based on the efficacy and safety data from the first phase, the investigators will optimize the trial design (primarily including the primary endpoint and sample size calculation) to evaluate the efficacy and safety of nanocrystalline megestrol acetate compared with dexamethasone, each combined with a 5-HT3 receptor antagonist, for the prevention of nausea and vomiting caused by moderately emetogenic chemotherapy drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, no gender restrictions;
2. Histologically or cytologically confirmed locally advanced/recurrent or metastatic gastric adenocarcinoma that is unresectable for curative treatment;
3. No prior exposure to any chemotherapy drugs (anticancer drugs not used for cancer treatment, or intravesical instillation therapy for bladder cancer is not considered chemotherapy);
4. First-line treatment planned to include a moderately emetogenic chemotherapy agent, specifically a PD-1 inhibitor (Tislelizumab is recommended), in combination with the CAPOX chemotherapy regimen for anticancer therapy;
5. Expected survival ≥ 6 months;
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
7. Good organ function, meeting the following criteria:

   1. Neutrophil count ≥ 1.5 × 10⁹/L;
   2. Hemoglobin ≥ 90 g/L;
   3. Platelet count ≥ 100 × 10⁹/L;
   4. Total bilirubin ≤ 1.5 × ULN;
   5. In patients without known liver metastases, aspartate aminotransferase ≤ 2.5 × ULN and/or alanine aminotransferase ≤ 2.5 × ULN (for patients with liver metastases, this may be relaxed to ≤ 5 × ULN);
   6. Serum creatinine ≤ 1.5 × ULN and creatinine clearance ≥ 50 mL/min;
   7. Electrocardiogram: QTc ≤ 450 ms (male), QTc ≤ 470 ms (female);
   8. Echocardiogram: LVEF (left ventricular ejection fraction) ≥ 50%;
8. Female participants of childbearing potential, as well as male participants whose partners are of childbearing potential, must use an effective method of contraception from the time of signing the informed consent form until 6 months after the last dose; female participants of childbearing potential must have a negative blood pregnancy test within 72 hours prior to randomization; and must not be breastfeeding;
9. Clearly understand and voluntarily participate in this study, and sign the informed consent form personally.

Exclusion Criteria:

1. Received abdominal (including the diaphragmatic plane and below) or pelvic radiotherapy within 7 days prior to enrollment, or plans to receive such radiotherapy between days 1 and 8 of treatment;
2. Plans to administer other chemotherapy drugs with moderate to high emetogenic potential between days 2 and 8 following the first day of chemotherapy;
3. History of venous thromboembolic disease within the past 6 months;
4. Use of medications with potential antiemetic effects within 2 days prior to enrollment: 5-HT3 receptor antagonists (e.g., ondansetron), phenothiazines (e.g., chlorpromazine), butyrophenones (e.g., haloperidol), benzamides (e.g., metoclopramide), domperidone, cannabinoids, traditional Chinese medicines with potential antiemetic effects, scopolamine, or secobarbital;
5. Initiation of benzodiazepine or opioid therapy within 2 days prior to enrollment (excluding zolpidem, temazepam, or midazolam taken alone daily);
6. Initiation of morphine use within 7 days prior to enrollment (excluding those on a stable dose);
7. Received systemic corticosteroid therapy (including but not limited to dexamethasone, hydrocortisone, methylprednisolone, or prednisolone) or sedating antihistamines (e.g., diphenhydramine) within 7 days prior to enrollment (Note:

   Single-dose corticosteroids for contrast medium allergy prevention, as well as local administration or inhalation, are permitted);
8. Use of palonosetron within 14 days prior to enrollment;
9. Use of NK-1 receptor antagonists within 28 days prior to enrollment;
10. Use of specific CYP3A4 substrates (terfenadine, cisapride, astemizole) or CYP3A4 inhibitors (e.g., ritonavir, clarithromycin, ketoconazole, or itraconazole, diltiazem, etc.), use of strong CYP3A4 inducers (e.g., phenobarbital, rifampin, phenytoin, and carbamazepine) within 28 days prior to enrollment, or use of specific CYP2D6 substrates (e.g., thioridazine, pimozide) within 28 days prior to enrollment;
11. Vomiting and/or nausea within 24 hours prior to enrollment;
12. Symptomatic brain metastases or any symptoms suggestive of brain metastases or intracranial hypertension;
13. Uncontrolled serous effusion, including pleural effusion, ascites, or pericardial effusion (patients who have achieved control through treatment and have been stable for ≥2 weeks may be included);
14. Severe cardiovascular disease within 3 months prior to enrollment, including but not limited to acute myocardial infarction, unstable angina, significant valvular or pericardial disease, history of ventricular tachycardia, symptomatic chronic heart failure (New York Heart Association [NYHA] Class II to IV), or history of severe cardiac conduction abnormalities (e.g., torsades de pointes);
15. Uncontrolled hypertension prior to enrollment (two consecutive resting systolic blood pressure readings ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg);
16. Active hepatitis B (HBV DNA ≥ 2000 IU/mL or 10⁴ copies/mL), active hepatitis C (HCV-Ab positive and HCV-RNA ≥ upper limit of normal), acquired immunodeficiency syndrome (AIDS) or HIV-positive, or syphilis-positive;
17. Concurrent conditions that preclude the use of dexamethasone, such as active infections (e.g., pneumonia) or any uncontrolled conditions (e.g., diabetic ketoacidosis, gastrointestinal obstruction, etc.);
18. Known contraindications to NK-1 receptor antagonists, 5-HT3 receptor antagonists, or dexamethasone;
19. Participation in other clinical trials within 30 days prior to enrollment (as determined by the use of study drugs);
20. Subjects deemed by the investigator to have other conditions that make them unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients without nausea during the entire period (Day 1-Day 21) after the start of chemotherapy drug administration in the first chemotherapy cycle. | the entire period (Day 1-Day 21) after the start of chemotherapy drug administration in the first chemotherapy cycle.